CLINICAL TRIAL: NCT01163955
Title: A Postural Analysis of Children Playing Video Games Sitting on the Floor vs. Sitting in a Chair: A Randomised Controlled Trial
Brief Title: A Postural Study Comparing Sitting on the Floor Versus Sitting in a Chair While Playing Video Games.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glinn and Giordano Physical Therapy (Other)
Responsible Party: Principal Investigator, Willam Brian Monroe, Physical Therapist, Glinn and Giordano Physical Therapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Protocol 10-90
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Results first posted 2011-09-30 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Scoliosis
Keywords: Posture analysis; Video gaming; Forward Head Position; Rounded Shoulder Position; Spine Posture
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitting in a chair (Other): Sitting in a chair with back support and feet flat on the ground
  Interventions: Other: Time to fatigue
- Sitting on the Floor (Other): Sitting on the floor without back support, crossed leg style
  Interventions: Other: Time to fatigue

INTERVENTIONS:
Other: Time to fatigue — 5 minutes while playing video games

SUMMARY:
To determine if sitting in a chair or sitting on the floor lends itself to better posture while playing video games.

DETAILED DESCRIPTION:
Upon completion of the parental consent form, each test subject will be instructed to flip a two-sided coin to determine the sitting position of the test subject. If the flip reveals a "heads", the child will be instructed to sit in a chair; chairs will be appropriately sized to allow the child to rest his/her feet on the ground. If the flip reveals a "tails", the child will be instructed to sit on a small carpet piece that measures 2-feet by 2-feet. Each test subject will be taken to their gaming station which will sit approximately 8 feet away from a 55-inch flat screen television that will be on a 30-inch table and handed a wireless controller. Two gaming stations will be available with one featuring the game Lego Batman and the other featuring Lego Indiana Jones with both gaming stations testing simultaneously. The test subjects will be told they can play for 5 minutes with a Physical Therapist at each station to monitor and record the test subjects' positioning.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish Speaking

Exclusion Criteria:

* Non-english or non-spanish speaking

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Monroe, DPT, OCS, Principal Investigator — Glinn and Giordano Physical Therapy; Erin P Pandol, MPT, OCS, Principal Investigator — Glinn and Giordano Physical Therapy
Locations (1):
- Best Buy Electronics, Bakersfield, California, United States

REFERENCES:
- See also: Related Info — http://www.ggphysicaltherapy.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Random recruitment at a Best Buy store. Flip of a coin decided the sitting position for the test
Pre-assignment Details: Some children were excluded from the final results because they sat on their glut max and kneeled alternating throughout the test.
Groups:
- Sitting in a Chair 5 Minutes: Sitting in a chair with back support and feet flat on the ground
- Sitting on the Floor 5 Minutes: Sitting on the floor without back support, crossed leg style
Period: Overall Study
Arm/Group | Sitting in a Chair 5 Minutes | Sitting on the Floor 5 Minutes
Started | 26 | 30
Completed | 26 | 26
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitting in a Chair 5 Minutes | Sitting on the Floor 5 Minutes | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 30 | 56
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.7 (2.5) | 8.8 (2.5) | 8.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  United States | 26 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: Posture Control of Head Position, Shoulder Position and Back Position
Description: Forward Head Position (FHP), Rounded Shoulder Position (RSP), and Thoracic spine (T/s)-Lumbar spine (L/s) positions were scored. Subscale scores of 0-3 for each FHP, RSP, and T/s L/s position were obtained. Score 0 was a perfect posture score, Score 1 was 0-1 inches out of alignment. Score 2 was 1-2 inches out of alignment. Score 3 was 2-3 inches out of alignment. Subscale scores were combined for a total score with a minimum value of 0 and a maximum value of 9. 0 being a perfect posture score, 9 being the worst postural score.
Time Frame: 5 minute
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Postural Score Sitting on Floor After 5 Minutes: Children sat on the floor for five minutes while playing a video game. No intervention (verbal or non-verbal) was given to them.
- Postural Score Sitting in a Chair After 5 Minutes: Children sat in a chair for five minutes while playing a video game. No intervention (verbal or non-verbal) was given to them.
Arm/Group | Postural Score Sitting on Floor After 5 Minutes | Postural Score Sitting in a Chair After 5 Minutes
Number analyzed (Participants) | 26 | 26
scores on a scale | 5.5 [2 to 9] | 2.8 [0 to 8]
Statistical Analysis 1: Comparison: Postural Score Sitting on Floor After 5 Minutes; Start total score at 0 minutes is being compared to the end total score at 5 minutes while sitting in the floor; Test type: Superiority or Other; p < .0005, t-test, 2 sided; DF=50; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [0 to 9], Standard Deviation 1.92
Statistical Analysis 2: Comparison: Postural Score Sitting in a Chair After 5 Minutes; Start total score at 0 minutes is being compared to the end total score at 5 minutes while sitting in a chair; Test type: Superiority or Other; p < .0005, t-test, 2 sided; DF=50; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [0 to 9], Standard Deviation 1.99

ADVERSE EVENTS:
Arm/Group | Sitting in a Chair 5 Minutes | Sitting on the Floor 5 Minutes
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes